CLINICAL TRIAL: NCT01845909
Title: Sudden Cardiac Death: Evaluation of a New Strategy to Identify Young Adults at Risk
Brief Title: Sudden Cardiac Death - Screening Of Risk Factors
Acronym: SCD-SOS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Coimbra (Other)
Collaborators: Unidade Local de Saúde de Coimbra, EPE (Other); Administração Regional de Saúde do Centro (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Rui Providência, M.D. M.Sc., University of Coimbra
Other Study IDs: SCD-SOS
Record Dates: First submitted 2013-04-27; First posted 2013-05-03 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Sudden Cardiac Death; Cardiomyopathies; Channelopathies
Keywords: Sudden cardiac death; Young adults; Cardiac Disease; Arrhythmia; Sports
MeSH Terms: conditions — Death, Sudden, Cardiac; Cardiomyopathies; Channelopathies; Heart Diseases; Arrhythmias, Cardiac | interventions — epicatechin gallate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- young adults - Central region of Portugal
  Interventions: Other: ECG and survey screening

INTERVENTIONS:
Other: ECG and survey screening

SUMMARY:
The investigators have created a way of quickly collecting information in a large scale young population regarding the presence of some severity indicators that may allow us to classify them into: seemingly "low risk" and possible "elevated risk" for the presence of heart disease. It would have to be a short questionnaire, in order to receive a great adherence but that could simultaneously provide precise information, with an adequate description of symptoms and warning signs, in a way that a triage in the young adult population could be performed in the general young adult population in order to select individuals with an indication for personalized clinical evaluation and possible need of complementary diagnostic means. Based on this premise the investigators have developed a fast-response questionnaire named the Sudden Cardiac Death Screening Of risk factorS (SCD-SOS). This questionnaire has already been tested in a population of approximately 1500 young adults, and some changes have been introduced in order to refine its performance.

To best of the investigators knowledge, there are no large scale European surveys estimating the prevalence of cardiac disease and associated clinical symptoms in a non-selected (non-athlete) population of this age group.

Purpose: To screen a young adult population from central regional of Portugal for heart disease possibly associated to a high risk of Sudden Cardiac Death (SCD).

To determine the national prevalence of clinical symptoms of heart disease and of heart disease with increased risk for SCD in this age group.

To detect young adults in risk of SCD and with an indication for evaluation by a cardiologist, and possible need of:

* medical treatment
* electrophysiologic (EP) study and percutaneous ablation
* an implantable cardiovertor defibrillator
* a pacemaker
* other type of specialized cardiac intervention

ELIGIBILITY:
Inclusion Criteria:

* 12 to 40 years of age
* Providing an informed consent

Exclusion Criteria:

* Failure to meet any of the aforementioned inclusion criteria

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Recruitment will include mainly university students but also young adults involved in sport practice (professional, semi-professional and amateur athletes) or in other activities (sales, industry, etc). This way, the places for sample collection will the university departments or technical schools, students associations and other places that gather university students, shopping centers, gyms, sports venues, factories in the city surroundings. Information collection in these places will be performed under the authorization of proper entities.
Sampling Method: Non-Probability Sample
Enrollment: 15351 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Type 1 electrocardiogram | baseline
  Presence of ECG changes suggestive of cardiac disease associated with an increased risk of sudden cardiac death. Definition present in:
  Corrado D et al. Recommendations for interpretation of 12-lead electrocardiogram in the athlete. Eur Heart J 2010;31:243-259
Clinical History - Red Flag | Baseline
  Presence of answers concerning symptoms or past family history that are known to be associated with increased risk of sudden cardiac death:
  e.g. effort syncope, syncope with fast palpitations prodrome, know high-risk cardiac disease, history of sudden cardiac death in first or second degree relative
all-cause mortality | First 20 years after enrollement
  occurrence of death of any cause in the participant
Cardiovascular death | First 20 years after enrollement
  Occurrence of death of cardiovascular etiology during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Providência, M.D. M.Sc., Study Chair — Coimbra's Hospital Centre and University; Faculty of Medicine, University of Coimbra, Portugal
Locations (1):
- Unidade Móvel - Tenda de Rastreio - SCDSOS, Coimbra, State..., Portugal